CLINICAL TRIAL: NCT05800678
Title: Comparison of Cross-sectional Area of Pubovisceral Muscle in Nulliparous and Primiparous Women
Brief Title: Cross-sectional Area of Pubovisceral Muscle in Nulliparous and Primiparous Women
Status: Completed | Type: Observational
Sponsor: Institute for the Care of Mother and Child, Prague, Czech Republic (Other)
Responsible Party: Principal Investigator, Katarina Ivankova, Principal investigator, Institute for the Care of Mother and Child, Prague, Czech Republic
Other Study IDs: UPMDPrague2021/28_1/2
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Pelvic Floor Disorders
Keywords: magnetic resonance imaging; levator ani muscle; denervation
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- nulliparous: inclusion: reproductive age
  exclusion: history of gynecological surgery or disorder with possible impact on pelvic floor
- primiparous: Inclusion: reproductive age, vaginal birth
  exclusion:
  * history of gynecological surgery or disorder with possible impact on pelvic floor
  * assisted vaginal delivery (forceps, vaccumextraction)
  * labour induction
  * pregnancy-related disorders
  * perineal tear grade III-IV (women with episiotomy were included)
  * suspicion of LAM avulsion by ultrasound or palpation
  * Oxford score 4 or 5 after delivery

SUMMARY:
Pelvic-floor disorders (PFD), including pelvic organ prolapse, urinary and fecal incontinence, decrease quality of life of every fourth women. 1 The main known risk factor for PFD is vaginal delivery 2,3 causing pelvic floor muscle avulsion, ischemia or denervation.4 Ultrasound (US) and magnetic resonance imaging (MRI) are frequently used to investigate structural changes in pelvic floor muscles. The investigators aimed to focus on structural changes (atrophy) caused by muscle denervation. 5 The pubovisceral muscle (PVM) is the part of the levator ani muscle (LAM) which is most frequently injured and it is thought to be possibly denervated by overstretching 6 Recently, the most precise measurement of PVM cross-sectional area was performed by the group of DeLancey. 7 In our study, the investigators aimed to describe which are the normal values of PVM volume in nulliparous women. The investigators performed a measurement of PVM volume in women after the first vaginal delivery.

The investigators hypothesized that there will be a decrease of the cross-sectional area of the PVM developed after denervation trauma.

DETAILED DESCRIPTION:
Two groups of women were recruited. First, the nulliparous group served as a control. The second group was women after their first vaginal delivery. Personal characteristics, anamnestic and delivery data were collected, and clinical examination, ultrasound (US) and magnetic resonance imaging (MRI) was performed. The number of women to reach significance in the study was 40/per group. The investigators did not expect a transfer of patients between the two groups. Volunteers were recruited from a general gynecological outpatient clinic. They were thoroughly informed and informed consent was provided.

In nulliparous women, all examinations (clinical, US, MRI) were performed only once. In women after vaginal delivery, first US was performed within 72h after childbirth, in order to detect LAM avulsion and exclude these women. In women without avulsion, 6 weeks after delivery, during a general postpartum checkup, the clinical evaluation of pelvic floor muscle contraction was performed. In those where the score is 0-3 the 3D US was performed to confirm no change of hiatal area during contraction. Those scans were recorded as investigated data. Those women underwent MRI within 4 months US images were obtained with a GE Voluson E10 system (General Electric Healthcare, Chicago, IL) by one investigator. US data acquisition was performed translabial as already described.9 Volumes were acquired at rest, during Valsalva and contraction. From acquired volume was assessed PVM avulsion, size of urogenital hiatus. Decrease of hiatal area at contraction proves muscle function. The assessment of US scans was performed off-line at axial plane using the 4D View v 2.1-5.0 software (GE Medical Systems) by two investigators blinded against all clinical data. MRI images were obtained with a 3-T scanner (AchievaTM, Philips Healthcare). MRI included coronal, axial, and sagittal proton density-weighted sequences performed at rest, Valsalva and contraction. Primary outcome evaluated by MRI will be the cross-sectional area of the PVM. The precise MRI technique was already defined by the group of DeLancey and is in detail described in recent publication.7 Evaluation was performed off-line by two investigators blinded against all clinical data using ImageJ software. Intra- and interobserver variability was calculated.

ELIGIBILITY:
Inclusion Criteria:

* reproductive age
* vaginal birth

Exclusion Criteria:

* history of gynecological surgery or disorder with possible impact on pelvic floor
* forceps, vaccumextraction)
* labour induction
* pregnancy-related disorders
* perineal tear grade III-IV (women with episiotomy were included)
* suspicion of LAM avulsion by ultrasound or palpation
* Oxford score 4 or 5 after delivery

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients of the Institute for the care of mother and child, Prague CZ
  * outpatient clinic
  * delivery ward and postpartum care unit
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
cross-sectional area of pubovisceral muscle | in nulliparous group measurements performed imediately after MRI. In primiparous group the MRI was performed within 3-6 months after delivery
  The PVM CSA was measured as previously described by Masteling et al.. Briefly, the MR images were imported into 3D Slicer, where slices containing the volume of interest were identified in a plane perpendicular to the muscle direction. To identify a plane perpendicular to the PVM, the PVM fibres direction was first established between origin and insertion, namely the inner surface of the pubic bone and its insertion into the perineal structures. In the coronal plane perpendicular to the muscle direction, the boundaries of the PVM were identified and images of this region were taken. The captured images were then exported into ImageJ for measurement of CSA.

CONTACTS AND LOCATIONS:
Overall Officials: Lucie Hájková Hympánová, PhD, Principal Investigator — Ústav pro péči o matku a dítě, Praha, CZ
Locations (1):
- Institute for mother and child care, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nygaard I, Barber MD, Burgio KL, Kenton K, Meikle S, Schaffer J, Spino C, Whitehead WE, Wu J, Brody DJ; Pelvic Floor Disorders Network. Prevalence of symptomatic pelvic floor disorders in US women. JAMA. 2008 Sep 17;300(11):1311-6. doi: 10.1001/jama.300.11.1311. PMID 18799443
- [Background] DeLancey JO. The hidden epidemic of pelvic floor dysfunction: achievable goals for improved prevention and treatment. Am J Obstet Gynecol. 2005 May;192(5):1488-95. doi: 10.1016/j.ajog.2005.02.028. PMID 15902147
- [Background] MacArthur C, Wilson D, Herbison P, Lancashire RJ, Hagen S, Toozs-Hobson P, Dean N, Glazener C; Prolong study group. Urinary incontinence persisting after childbirth: extent, delivery history, and effects in a 12-year longitudinal cohort study. BJOG. 2016 May;123(6):1022-9. doi: 10.1111/1471-0528.13395. Epub 2015 Apr 2. PMID 25846816
- [Background] Weidner AC, Jamison MG, Branham V, South MM, Borawski KM, Romero AA. Neuropathic injury to the levator ani occurs in 1 in 4 primiparous women. Am J Obstet Gynecol. 2006 Dec;195(6):1851-6. doi: 10.1016/j.ajog.2006.06.062. PMID 17132486
- [Background] Carlson BM. The Denervated Muscle: 45 years later. Neurol Res. 2008 Mar;30(2):119-22. doi: 10.1179/174313208X281127. PMID 18397601
- [Background] DeLancey JO, Sorensen HC, Lewicky-Gaupp C, Smith TM. Comparison of the puborectal muscle on MRI in women with POP and levator ani defects with those with normal support and no defect. Int Urogynecol J. 2012 Jan;23(1):73-7. doi: 10.1007/s00192-011-1527-8. Epub 2011 Aug 6. PMID 21822711
- [Background] Masteling M, Ashton-Miller JA, DeLancey JOL. Technique development and measurement of cross-sectional area of the pubovisceral muscle on MRI scans of living women. Int Urogynecol J. 2019 Aug;30(8):1305-1312. doi: 10.1007/s00192-018-3704-5. Epub 2018 Jul 5. PMID 29974138